CLINICAL TRIAL: NCT06731283
Title: Evaluation of Serological Markers of Vitiligo Activity
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0610
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Vitiligo
Keywords: biomarker; vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vitiligo: Patients diagnosed with vitiligo
- Controls: Patients that do not have vitiligo

SUMMARY:
The goal of this case-control study is to evaluate the possible applicability of CXCL10, CXCL9, CCL20, and homocysteine as biomarkers of disease activity in vitiligo patients and to compare the levels of these markers with those in healthy controls.

DETAILED DESCRIPTION:
The diagnosis and prognosis assessment in patients with vitiligo are essentially clinical. There are still no validated and established serological markers to objectively assist in defining disease activity. Objective: To evaluate the potential use of the biomarkers CXCL9, CXCL10, CCL20, S100B, and homocysteine to identify disease activity in vitiligo, comparing their values with controls. Methods: A case-control study using previously collected peripheral blood samples from patients aged 18 years or older with a diagnosis of vitiligo and from controls without the disease. The project was approved by the institution's ethics committee. Tests were conducted using ELISA and Luminex kits to measure CXCL9, CXCL10, CCL20, and S100B. For homocysteine, the chemiluminescence method was used.

ELIGIBILITY:
Inclusion Criteria:

* Vitiligo
* Older than 18 years

Exclusion Criteria:

* Not having diagnosis of vitiligo
* Less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Dermatology Department of Hospital de Clínicas de Porto Alegre
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Biomarkers levels | through study completion, an average of 2 year
  Assessment of the biomarkers levels in vitiligo group and group control

CONTACTS AND LOCATIONS:
Overall Officials: Tania Cestari, Professor, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No